CLINICAL TRIAL: NCT02197897
Title: Phase II Trial of Estrogen Receptor Targeted Treatment of Non-Muscle Invasive Bladder Cancer With Tamoxifen.
Brief Title: Evaluation the Treatment of Tamoxifen of Low/Intermediate Risk Bladder Tumors
Acronym: BCTamoxifen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guilherme Godoy, Guilherme Godoy, M.D., Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-25233; K23CA160664 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Bladder Cancer
Keywords: Tamoxifen citrate; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tamoxifen (Experimental): As a single-arm study (single group assignment), Tamoxifen citrate will be given to all patients at a 20mg/day dose for 12 weeks using a marker-lesion study design.
  Interventions: Drug: Tamoxifen Citrate

INTERVENTIONS:
Drug: Tamoxifen Citrate — Single-center, two-stage phase-II clinical trial (Simon design)
  Other Names: Nolvadex

SUMMARY:
Evaluate the treatment of tamoxifen of low/intermediate-risk bladder tumors

DETAILED DESCRIPTION:
Patients with primary or recurrent low/intermediate-risk papillary urothelial carcinoma of the bladder will undergo resection of all but one marker lesion, measuring at least 6mm but no greater than 10mm, and biopsy of normal-appearing mucosa. Patients with a solitary tumor will undergo only biopsy prior to treatment. A 2mm cold cup biopsy of the marker lesion will always be performed to rule out a potential high-grade lesion and for assessment of pretreatment immunohistochemistry expression levels of ERα, ERβ1, Ki-67 (proliferation marker) and TUNEL (apoptosis marker). If there are multiple tumors, all lesions, except the marker lesion will be resected and sent for analysis. These patients will not receive single immediate post-operative intravesical instillation of mitomycin-C. They will then undergo a 12-week course of treatment with tamoxifen administered as a single daily oral dose of 20mg. At the completion of therapy, patients will undergo resection of the marker lesion (or biopsy of the tumor bed, if a complete response is observed) and biopsy of normal-appearing bladder mucosa again. Toxicity evaluations will be performed at the beginning (day 3), midway (week 6), and at completion of treatment (week 12), prior to resection of the marker lesion. A final assessment for toxicity will also be performed 30 days after completion of therapy as well as a second definitive resection of the marker lesion. Urine samples will be obtained with the index tumor in place (marker lesion), and after completion of treatment, at the time of definitive transurethral resection of the index tumor, as part of the standard clinical care of these patients, and at the discretion of the surgeon for assessment of urinary cytology. The urine samples will not be utilized for the research study. All normal-appearing bladder biopsies (pre and post-treatment), the additional tumors (in case of multiple lesions), and the definitive resection of the marker lesion (in the absence of response to therapy) will provide sufficient material for immunohistochemistry assessment of the expression levels of ERα, ERβ-1, ERβ-2, ERβ-5, Ki-67, and TUNEL, and also for RT-qPCR for mRNA analyses of ERα, ERβ-1, ERβ-2, and ERβ-5. The pretreatment biopsy of the marker lesion will be performed with a smaller biopsy forceps and will provide limited material, sufficient only for immunohistochemistry assessment of the expression levels of ERα, ERβ-1, Ki-67, and TUNEL.

ELIGIBILITY:
Inclusion Criteria:

Males and females age 21 or older. Histologic evidence of urothelial carcinoma of the bladder. Low/Intermediate-risk papillary urothelial carcinoma of the bladder, at initial occurrence or recurrent with >6 months interval free of disease.

Patients with multifocal tumors must have resectable lesions. Patients may be treatment-naïve or have failed 1 previous regimen of intravesical therapy.

At least one endoscopically measurable tumor 6 - 10mm in diameter. Adequate hepatic and renal function. Patient or authorized proxy needs to have signed the informed consent form.

-

Exclusion Criteria:

Patients with sessile appearing tumors, which may be invasive or high-grade. Diagnosis of urothelial carcinoma involving the prostatic urethra or upper urinary tract.

Plans for pelvic radiation while participating in the study. Concurrent use of warfarin, heparin, or chronic use of NSAIDs, including aspirin (other than cardioprotective doses of 80mg daily) within 30 days prior to registration or during the trial.

Concurrent use of selective serotonin reuptake inhibitors or aromatase inhibitors.

Chronic or acute renal or hepatic disorder or any other condition, medical or psychological that, in the opinion of the investigator, could jeopardize the subject's safe participation.

Any other investigational drug within 30 days prior to registration and during the study.

Women Exclusion Pregnant or lactating women. Personal history of endometrial cancer or any abnormal uterine bleeding. Previous or concurrent treatment with SERM and/or hormonal replacement therapy within 3 months of the study.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Godoy, M.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Harris Health System, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be identified from the Scott Department of Urology (SDU) and Affiliated Institutions.Patients will be informed verbally and in writing about the study, procedures involved. They will be given adequate opportunity to read it and discuss with family before it is signed. Participation in this study will last about 4 months.
Period: Overall Study
Arm/Group | Tamoxifen
Started | 15
Completed | 14
Not Completed | 1
Not completed — not eligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tamoxifen
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Ethinicity: Asian | 1
  Race Ethinicity: Black | 2
  Race Ethinicity: White | 10

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Efficacy for Treatment of Low/Intermediate- Risk Bladder Tumors, Assessing for the Clinical Response of the Marker Lesion
Description: Evaluate the efficacy of tamoxifen for treatment of low/intermediate-risk bladder tumors, utilizing the RECIST criteria combined with the final biopsy of the marker lesion or the bed of the lesion in case of a complete response
Time Frame: 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tamoxifen
Number analyzed (Participants) | 14
Participants | 13

ADVERSE EVENTS:
Time Frame: Clinical toxicity evaluations (secondary aim 1d) were performed at the beginning (postoperative day 3), midway (postoperative week 6), and at completion of treatment (postoperative week 12), prior to the final resection of the marker lesion. A final assessment for toxicity was also performed 30 days after completion of therapy and definitive resection of the marker lesion.
Description: Toxicity events were recorded utilizing the Common Terminology Criteria for Adverse Events version 4.02 (CTCAE v4.02). Figure 1 illustrates the study linear chronogram schema.
Arm/Group | Tamoxifen
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen (N=13)
Hematuria (Blood and lymphatic system disorders) | 3 (3)
Urinary Tract Pain (Gastrointestinal disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolic event (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Non Cardiac Chest Pain (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Platelet Count decreased (Blood and lymphatic system disorders) | 2 (3)
Blood Bilirubin Increase (Blood and lymphatic system disorders) | 1 (1)
creatinine increase (Blood and lymphatic system disorders) | 1 (2)
Lymphocyte Count decrease (Blood and lymphatic system disorders) | 1 (2)
Hypocalcemia (Blood and lymphatic system disorders) | 2 (3)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (2)
Eye Disorders (Eye disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Erectile Dysfunction (General disorders) | 1 (1)
Dyspenia (General disorders) | 1 (2)
Rash Maculo- Papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02197897/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT02197897/Prot_SAP_001.pdf